CLINICAL TRIAL: NCT03142750
Title: Design of a Dressing for Gastrostomy Buttons in Pediatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-0063
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Gastrostomy Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Enrolled subjects (Experimental): There is only one arm to this study. The intervention includes providing one week supply of each of two gastrostomy tube dressing prototypes to try at home.
  Interventions: Device: Gastrostomy tube dressing

INTERVENTIONS:
Device: Gastrostomy tube dressing — Two types of dressings to secure gastrostomy tube in children

SUMMARY:
Gastrostomy tube (G-tube) complications, such as granulation tissue formation and tube dislodgements, are frequent causes of emergency department visits. The investigators have developed two G-tube dressing designs using commercially available materials and products to decrease the risk of G-tube related complications. The investigators aim in this study is to pilot two novel G-tube dressings in patients with pre-existing G-tubes to gain parental feedback on device designs, ease of use and G-tube stability in preparation for a final design and trial. Based on the feedback, further iterations will be developed and trialed in eligible study subjects.

DETAILED DESCRIPTION:
In order to address complications associated with gastrostomy buttons (G-buttons) or tubes (G-tubes) in children, the investigators developed two multi-component securement dressings. The purpose of this study is to try these dressings and obtain parental feedback.

This will involve survey using questionnaires before and after the use of two different G-tube dressings. Eligible patients will be identified by a nurse practitioner or attending surgeon. The researcher will obtain consent from the patient or their parents/legal guardian. The investigators will ask a series of questions regarding their current experience dressing and maintaining G-tube stomas. A week supply of each new prototype dressing will be provided to the patient or parent. Caregivers will be educated on the use of each dressing and will be given a number to call should they have any questions or concerns. The dressings will be changed daily and as needed. Once the patient is enrolled and provided with dressings, the investigators will perform a follow up telephone interview at one week to evaluate their experience and ensure they did not experience any adverse events. Caregivers will be given a second questionnaire to collect feedback on the dressings after two weeks either in person or over the telephone. They will be asked to choose their preferred dressing, provide feedback on advantages and disadvantages of each type and report adverse events. For inpatients, the investigators will obtain opinions from parents, patients, nurses and doctors. Photographs will be obtained at each outpatient visit or during the inpatient period for objective comparison.

Once more iterations are developed, they will undergo the same clinical trial process (involving 10-15 subjects).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pre-existing a G-tube
* Patients presenting to the G-tube or surgery clinic for G-tube replacement at Children's Hospital, Aurora, Colorado.
* Patients admitted to the hospital with a pre-existing G-tube for reasons unrelated to the G-tube will be eligible for the study if they have issues with the G-tube site.

Exclusion Criteria:

* Refusal to participate
* Those with other types of gastrostomy tubes (other than Mini Balloon Button)
* Those whose parents or legal guardians cannot be reached by telephone
* Prisoners
* Pregnant women
* Decisionally challenged subjects

Ages: 31 Days to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Moulton, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Saddle and Foam Gastronomy Tube Dressing: The intervention includes providing one week supply of each of two gastrostomy tube dressing prototypes to try at home.
  Gastrostomy tube dressing: Two types of dressings to secure gastrostomy tube in children
- Experimental: Gastronomy Tube Dressing Prototype: A third prototype gastronomy tube dressing will be created using the feedback collected from the first group of subjects about the Saddle and Foam dressings. A new group of participants will receive the prototype dressing.
Period: Overall Study
Arm/Group | Experimental: Saddle and Foam Gastronomy Tube Dressing | Experimental: Gastronomy Tube Dressing Prototype
Started | 14 | 10
Completed | 10 | 9
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Population: The initial 14 participants provided information for baseline measures. These participants trialed both the Foam and Saddle Gastrostomy Tube Dressings. Using the qualitative information provided from the first two experimental arms, a Third Dressing Prototype was created. A separate group of 10 participants trialed the third prototype.
Groups:
- Foam and Saddle Gastrostomy Tube Dressing: The intervention includes providing one week supply of each of two gastrostomy tube dressing prototypes to try at home.
  Gastrostomy tube dressing: Two types of dressings to secure gastrostomy tube in children
- Third Gastrostomy Tube Dressing Prototype: A third prototype gastronomy tube dressing will be created using the feedback collected from the first group of subjects about the Saddle and Foam dressings. A new group of participants will receive the prototype dressing.
- Total: Total of all reporting groups
Arm/Group | Foam and Saddle Gastrostomy Tube Dressing | Third Gastrostomy Tube Dressing Prototype | Total
Number analyzed (Participants) | 14 | 10 | 24
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 4 [1 to 7] | 4 [1 to 9] | 4 [1 to 9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 7 | 4 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 10 | 24
Newly placed gastrostomy button [Count of Participants; unit: Participants] | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Satisfied With Current Dressings
Description: Overall satisfaction of the current dressings used at baseline were assessed using a qualitative questionnaire. Questionnaires queried the level of agreement in the following aspects: overall satisfaction, ease of use, adequate level of security for the G-button, adherence to skin, ability to absorb leakage, cost, availability at drug store, allergenic potential and reusability. Answer choices to measure level of satisfaction were: strongly agree, agree, neutral, disagree, strongly disagree. Surveys also included open-ended questions about participant satisfaction. Survey responses were evaluated and determined to indicate "Satisfied" or "Not Satisfied" by the Investigators.This measurement reflects participants satisfaction with whatever dressing they were currently using at baseline, not with the study interventions to which they were assigned.
Time Frame: Baseline
Population: Only participants from the Foam Gastrostomy Tube Dressing and Saddle Gastrostomy Tube dressing completed this baseline measure. No participants from the Third Prototype group completed this baseline measure
Measure: Count of Participants; unit: Participants
Groups:
- Foam Gastronomy Tube Dressing: The intervention includes providing one week supply of each of two gastrostomy tube dressing prototypes to try at home.
  Gastrostomy tube dressing: Two types of dressings to secure gastrostomy tube in children
- Saddle Gastrostomy Tube Dressing: This group was given a 1 week supply of both the saddle and foam type gastrostomy tube dressing for trial at home.
- Third Prototype: Third prototype (silicone pod and flexible snap rings)
Arm/Group | Foam Gastronomy Tube Dressing | Saddle Gastrostomy Tube Dressing | Third Prototype
Number analyzed (Participants) | 8 | 8 | 0
Participants
  Number of participants satisfied with dressing | 3 | 3 |
  Number of participants not satisfied with dressing | 5 | 5 |

2. Primary Outcome: Number of Participants Satisfied With Experimental Dressings
Description: Overall satisfaction of the dressings when assessed using a qualitative questionnaire. Questionnaires queried the level of agreement in the following aspects: overall satisfaction, ease of use, adequate level of security for the G-button, ease of connecting and disconnecting the feeding tube, reduction in leakage, painless device removal, improvement in gastrostomy wound appearance, preference over the traditional dressing, and whether they would purchase the securement device if it was commercially available. Answer choices to measure level of satisfaction were: strongly agree, agree, neutral, disagree, strongly disagree. Surveys also included open-ended questions about participant satisfaction. Survey responses were evaluated and determined to indicate "Satisfied" or "Not Satisfied" by the Investigators.
Time Frame: 1 Week
Population: 4 subjects in the Saddle & Foam group and 1 in the Third Prototype did not complete the satisfaction surveys.
Measure: Count of Participants; unit: Participants
Groups:
- Foam Gastrostomy Tube Dressing: The intervention includes providing one week supply of each of two gastrostomy tube dressing prototypes to try at home.
  Gastrostomy tube dressing: Two types of dressings to secure gastrostomy tube in children
- Saddle Design Gastrostomy Dressing: The intervention includes providing a one week supply of each of the two gastrostomy tube dressings to ten participants to try at home.
Arm/Group | Foam Gastrostomy Tube Dressing | Saddle Design Gastrostomy Dressing | Third Prototype
Number analyzed (Participants) | 10 | 10 | 9
Participants
  Satisfied with dressing | 9 | 8 | 6
  Not satisfied with dressing | 1 | 2 | 3

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Dressing is not invasive. No risk for serious adverse event or mortality.
Groups:
- Foam Gastrostomy Dressing Prototype; Saddle Gastrostomy Dressing Prototype: The intervention includes providing one week supply of each of two gastrostomy tube dressing prototypes to try at home.
  Gastrostomy tube dressing: Two types of dressings to secure gastrostomy tube in children
  Only 10 participants completed follow up
- Third Gastrostomy Dressing Prototype: Using feedback from the Foam and Saddle groups a third Gastrostomy Dressing Prototype was created and trialed by a new group of participants
  Only 9 participants completed follow up
Arm/Group | Foam Gastrostomy Dressing Prototype | Saddle Gastrostomy Dressing Prototype | Third Gastrostomy Dressing Prototype
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/10
Other Adverse Events (participants affected / at risk) | 0/14 | 1/14 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Foam Gastrostomy Dressing Prototype (N=14) | Saddle Gastrostomy Dressing Prototype (N=14) | Third Gastrostomy Dressing Prototype (N=10)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Child developed small pinpoint rash under the dressing. It was noted after dressing was removed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/50/NCT03142750/Prot_000.pdf